CLINICAL TRIAL: NCT05361382
Title: Longitudinal Multicenter Head-to-Head Harmonization of Tau PET Tracers
Brief Title: Head-to-Head Harmonization of Tau Tracers in Alzheimer's Disease
Acronym: HEAD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tharick Pascoal (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Tharick Pascoal, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY22020056; R01AG073267 (NIH)
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease
Keywords: Tau PET; Neurofibrillary tangles; Alzheimer's disease; Tauopathies; Biomarkers
MeSH Terms: conditions — Alzheimer Disease; Tauopathies | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene; flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individuals across the aging and Alzheimer's disease (AD) spectrum (Experimental): All individuals enrolled into the HEAD study will undergo tau PET, amyloid-β PET, magnetic resonance imaging (MRI), detailed clinical and cognitive assessment, and a blood draw.
  Interventions: Drug: 18F-Flortaucipir radiopharmaceutical; Drug: 18F-MK-6240 radiopharmaceutical; Drug: Amyloid-β radiopharmaceutical (11C-PiB or 18F-Florbetaben or 18F-NAV-4694 or 18F-Flutemetamol)

INTERVENTIONS:
Drug: 18F-Flortaucipir radiopharmaceutical — Flortaucipir is a PET radiopharmaceutical that binds to tau neurofibrillary tangles. Participants will receive a bolus intravenous injection of approximately 10 millicuries of the radiopharmaceutical.
  Other Names: 18F-AV-1451, 18F-T807, Tauvid
Drug: 18F-MK-6240 radiopharmaceutical — MK-6240 is a PET radiopharmaceutical that binds to tau neurofibrillary tangles. Participants will receive a bolus intravenous injection of approximately 5 millicuries of the radiopharmaceutical.
Drug: Amyloid-β radiopharmaceutical (11C-PiB or 18F-Florbetaben or 18F-NAV-4694 or 18F-Flutemetamol) — The clinical sites will use either PiB, Florbetaben, Flutemetamol, or NAV-4694 as the amyloid-β PET radiopharmaceutical. The amyloid-β PET radiopharmaceutical binds to amyloid-β plaques.
  Participants will receive a bolus intravenous injection of approximately 15 millicuries of the PiB radiopharmaceutical.
  Participants will receive a bolus intravenous injection of approximately 8 millicuries of the Florbetaben or NAV-4694 radiopharmaceutical.
  Participants will receive a bolus intravenous injection of approximately 5 millicuries of the Flutemetamol radiopharmaceutical.

SUMMARY:
The purpose of this study is to compare/harmonize cross-sectional and longitudinal tau tangle measurements obtained with the tau PET radiopharmaceuticals Flortaucipir and MK-6240 to elucidate the advantages and caveats of their use in clinical trials/practice and provide parameters to integrate their estimates.

DETAILED DESCRIPTION:
This is a longitudinal, multi-site, non-randomized study in which the participants will undergo Flortaucipir and MK-6240 PET scans at baseline and approximately at 18-month follow-up. At each time point, participants will also have an amyloid-β PET scan, magnetic resonance imaging, detailed cognitive tests, and a blood draw for biomarker quantification. The main objectives of this study are standardizing tau PET tracers' outcomes and comparing their performance.

To accomplish our objectives, the investigators propose the following specific aims:

In Aim 1, investigators will standardize tau PET processing methods, convert the tracers to a common scale, compare associations with amyloid-β, atrophy, and cognition, and compare/harmonize Braak staging assessments between tau tracers using cross-sectional data.

In Aim 2, investigators will ascertain the optimal processing method for longitudinal analysis and compare longitudinal changes in tau accumulation obtained with the tau PET radiopharmaceuticals and their associations with changes in amyloid-β, atrophy, and cognition.

In Exploratory Aim 3, investigators will compare cross-sectional and longitudinal Flortaucipir and MK-6240 estimates with plasma phosphorylated tau concentrations.

This study will produce a benchmark dataset to develop methods for tau PET quantification and harmonization.

ELIGIBILITY:
Inclusion criteria:

* Have a study partner who will be able to provide an independent evaluation of functioning.
* Willing and capable of undergoing repeated MR/PET imaging.
* Fluent in a language approved by the coordinating center.
* At screening, must have no cognitive impairment, or meet criteria for single- or multiple-domain amnestic mild cognitive impairment or Alzheimer's disease dementia.

Exclusion criteria:

* Inability to provide informed consent by self or by proxy.
* Pregnant or breastfeeding women.
* Have any condition or are taking any medication that could increase the risk to the participant, limit the ability to tolerate or interfere with the results of the tests and procedures (in the opinion of the investigator).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional tau PET uptake values | 2 years from enrollment
  Compare/harmonize cross-sectional tau deposition measurements (standardized uptake value ratio (SUVR)) obtained with Flortaupicir and MK-6240.
Longitudinal change in tau PET uptake values over 18 months | 5 years from enrollment
  Compare/harmonize change in tau deposition measurements (standardized uptake value ratio (SUVR)) obtained with Flortaupicir and MK-6240 between baseline and 18-month follow-up assessments.

SECONDARY OUTCOMES:
Associations of tau PET uptake values with amyloid-β PET uptake values | 5 years from enrollment
  Compare the effect size of the associations of tau deposition measurements (standardized uptake value ratio (SUVR)) obtained with Flortaupicir and MK-6240 with amyloid-β deposition measurements (SUVR).
Associations of tau PET uptake values with measures of cognition | 5 years from enrollment
  Compare the effect size of the associations of tau deposition measurements (standardized uptake value ratio (SUVR)) obtained with Flortaupicir and MK-6240 with cognitive measures assessed from neuropsychological evaluation.
Associations of tau PET uptake values blood biomarkers | 5 years from enrollment
  Compare the effect size of the associations of tau deposition measurements (standardized uptake value ratio (SUVR)) obtained with Flortaupicir and MK-6240 with blood-based biomarkers of tau.

CONTACTS AND LOCATIONS:
Overall Officials: Tharick Pascoal, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (9):
- United States (7):
  - Lawrence Berkeley National Laboratory, Berkeley, California
  - University of California San Francisco, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Houston Methodist Neurological Institute, Houston, Texas
- McGill University, Montreal, Quebec, Canada
- Sant Pau Biomedical Research Institute, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data from this research will be shared with other researchers pursuant to the 02/26/2003 "NIH Final Statement on Sharing Research Data". To protect participants' rights and confidentiality, identifiers will be removed from the data before they are shared. The board of PIs has primary oversight of the HEAD study resource sharing plan and will review all issues related to internal and external requests for HEAD data. Raw PET and MR data will be uploaded by clinical sites after acquisitions, whereas processed PET and MR data will be uploaded after completion of the baseline visit and after completion of the 18-month follow-up visit. Demographics, results from cognitive tests, Aβ status, tau Braak staging, and plasma assay results will also be available through the LONI platform.
Time Frame: Data from baseline and follow-up assessments will be available for sharing after the completion of the respective study visits.
Access Criteria: Researchers will be able to download data upon request to the PIs. Data sharing requests will be overseen by the study and site PIs.
URL: http://www.loni.usc.edu/

DOCUMENTS (1):
  • Informed Consent Form (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT05361382/ICF_000.pdf